CLINICAL TRIAL: NCT03796416
Title: Obesity Study to Assess Induction of Labor With Balloon and Cytotec: a Randomized Control Trial
Brief Title: Obesity Study to Assess Induction of Labor
Acronym: Obtainable
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: in error
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Sarah Crimmins, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00077208
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- misoprostol (Active Comparator): Induction using misoprostol:
  Insert misoprostol 25 micrograms in the posterior fornix of the vagina digitally Repeat cervical exam every 4 hours
  Interventions: Drug: Misoprostol
- Misoprostol and foley bulb (Experimental): Induction using Foley balloon combined with misoprostol:
  A 26 French intracervical Foley balloon will be inserted above the internal os at the start of induction, inflated using 80cc of sterile water.
  If a Foley balloon is not able to be inserted at the time of starting induction of labor, misoprostol 25microgram can be inserted in the posterior fornix of the vagina and the misoprostol protocol followed.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — used at a rate of 25 mcg Q4hours for cervical ripening.

SUMMARY:
There are more and more pregnant women who are obese. It is very difficult for obese women to get into labor. That is why when women are obese, half are likely to need a Cesarean delivery(C-section). Unfortunately, C-sections are more dangerous for obese women. There may be a combination of issues that cause obese women to need C-sections. We believe one of those reasons is that the womb of obese women respond differently to medications and devices compared to non-obese women. There are commonly two ways to help women get into labor. One way is a medication called misoprostol. The second way is a device called Foley balloon. In most studies, both ways are equally effective in helping women get into labor. However, these studies included everyone, and didn't focus on obese women.

So far there are no studies in this area that focus only on obese women. Therefore we need to design this study to focus just on obese women and what is the best way to help them get into labor and avoid a C-section.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patient (BMI≥40kg/m2) at admission for induction of labor Speaks English Gestational age between 37and0 weeks and 41and6 weeks Cervical exam: dilation <4cm and Bishop score 6 or less Contractions < 2 per 10 minutes

Exclusion Criteria:

* History of cesarean delivery Maternal contraindications to labor Fetal contraindications to labor Maternal age <18yo Fetal growth restriction with abnormal umbilical artery Doppler indexes Cervical dilation ≥4cm or Bishop score ≥7 Contractions ≥3 per 10 minutes Non-reassuring fetal status Latex allergy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
achieving complete cervical dilation | 24 hours

IPD SHARING:
Plan to Share IPD: Undecided